CLINICAL TRIAL: NCT01273597
Title: Post-marketing Observational Study to Evaluate the Time to Achieving the Maintenance Dose of Paricalcitol i.v. in the Treatment of Chronic Kidney Disease (CKD) 5 Stage Patients With (Severe) Secondary Hyperparathyroidism in Hungary
Brief Title: Observational Study to Evaluate the Time to Achieving the Maintenance Dose of Zemplar® (Paricalcitol Injection) in the Treatment of Patients Suffering From End-stage Renal Disease and Severe Over-reactivity of the Parathyroid Glands
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Planimeter Ltd (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-644
Record Dates: First submitted 2010-11-22; First posted 2011-01-10 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Parathyroid hormone,Kidney failure, chronic,Hyperparathyroidism, secondary
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End-stage kidney disease with secondary hyperparathyroidism: Participants with chronic kidney disease (CKD) stage 5 receiving haemodialysis with a diagnosis of secondary hyperparathyroidism (SHPT)

SUMMARY:
This observational study will evaluate the clinical benefit of Zemplar (paricalcitol injection) in daily routine practice in end-stage renal disease patients with severe over-reactivity of parathyroid glands. Participants will be followed for 6 months. Data will be collected from participants initiated on Zemplar therapy according to standard of care. The time to achieving the maintenance dose of Zemplar (paricalcitol injection), the proportion of participants achieving target parathyroid hormone levels, and prevalence of elevated serum calcium and phosphate levels will be evaluated.

DETAILED DESCRIPTION:
Prospective data collection started at initial dosing with Zemplar (paricalcitol injection) and ended up to 6 months later. If available, retrospective data on vitamin D treatment as well as on the incidence of hypercalcaemia and hyperphosphataemia in the 6 months leading up to paricalcitol treatment were also collected. Eight visits were planned for documentation of prospective data. In accordance with the non-interventional character of the study, only diagnostic and monitoring procedures were applied which are part of the routine medical care of secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

Based on the current Hungarian Summary of Product Characteristics for Zemplar (paricalcitol injection), the patient is entitled to treatment with paricalcitol injection and:

1. ≥ 18 years of age,
2. Willing to sign the patient information and informed consent form,
3. Chronic kidney disease (CKD) stage 5 patient receiving haemodialysis with a diagnosis of secondary hyperparathyroidism (SHPT), whose intact parathyroid hormone (iPTH) level is:

   * between 500-800 pg/mL with at least two abruption of conventional vitamin D therapy due to elevated serum calcium level (i.e. > 2.4 mmol/L) in the medical history, or
   * higher than 800 pg/mL and parathyroidectomy is contraindicated.
4. The patient is planned to receive paricalcitol treatment independently from his/her participation in this study.

Exclusion Criteria:

Patients cannot be enrolled in the study if any of the following exclusion criteria apply:

1. The patient is already treated with Zemplar (paricalcitol injection),
2. Any contraindication exists as stated in the current Hungarian Summary of Product Characteristics for Zemplar (paricalcitol injection),
3. Patients who decline to participate in the study or decline to sign the patient information/informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 5 chronic kidney disease patients treated in haemodialysis centers in Hungary
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Schnaider, Study Director — AbbVie (prior sponsor, Abbott)
Locations (11):
- Hungary (11):
  - Site Reference ID/Investigator# 46593, Budapest
  - Site Reference ID/Investigator# 46585, Budapest
  - Site Reference ID/Investigator# 46594, Debrecen
  - Site Reference ID/Investigator# 47722, Győr
  - Site Reference ID/Investigator# 46592, Karcag
  - Site Reference ID/Investigator# 58644, Karcag
  - Site Reference ID/Investigator# 46595, Miskolc
  - Site Reference ID/Investigator# 46588, Nyíregyháza
  - Site Reference ID/Investigator# 46597, Pécs
  - Site Reference ID/Investigator# 46590, Szombathely
  - Site Reference ID/Investigator# 46591, Veszprém

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Started | 60
Completed | 52
Not Completed | 8
Not completed — Adverse Event | 5
Not completed — Underwent Kidney Transplantation | 2
Not completed — Reason Not Reported | 1

BASELINE CHARACTERISTICS:
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 60
Age Continuous [Mean (Full Range); unit: years] | 57.7 [31 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 29
Region of Enrollment [Number; unit: participants]
  Hungary | 60

OUTCOME MEASURES:

1. Primary Outcome: Time (in Weeks) From Treatment Initiation to Achieving Maintenance Dose of Zemplar (Paricalcitol Injection)
Description: Maintenance dose is defined as weekly dose of paricalcitol that results in at least 2 consecutive intact parathyroid hormone (iPTH) values within the target therapeutic range of 150 - 300 pg/mL, corresponding to 15.9 - 31.8 pmol/L.
Time Frame: 6 months
Population: Participants who achieved maintenance dose of Zemplar (paricalcitol injection)
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 16
weeks | 12.2 (7.6)

2. Secondary Outcome: Number of Participants Achieving Target Intact Parathyroid Hormone (iPTH) Levels at Month 6
Description: Target intact parathyroid hormone (iPTH) values were within the target therapeutic range of 150 - 300 pg/mL, corresponding to 15.9 - 31.8 pmol/L.
Time Frame: 6 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 60
participants | 14

3. Secondary Outcome: Country-Specific Data on the Usage of Medication Affecting Calcium (Ca) Balance
Description: If available, data on vitamin D treatment (those who received vitamin D supplement products from Anatomical Therapeutic Chemical [ATC] group A11CC [vitamin D and analogues]) in the 6 months leading up to paricalcitol treatment and during 6 months of paricalcitol treatment were also collected.
Time Frame: 6 months prior to start of study through 6 months of treatment
Population: This outcome measure was not analyzed due to lack of data.
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 0

4. Secondary Outcome: Country-Specific Data on the Usage of Medication Affecting Phosphorus (P) Balance
Description: If available, data on the use of phosphate binders (those who received calcium-based phosphate binders or sevelamer/lanthanum) in the 6 months leading up to paricalcitol treatment and during 6 months of paricalcitol treatment were also collected.
Time Frame: 6 months prior to start of study through 6 months of treatment
Population: This outcome measure was not analyzed due to lack of data.
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 0

5. Secondary Outcome: Country-Specific Data on the Usage of Medication Affecting Secondary Hyperparathyroidism
Description: If available, data on the use of medication affecting secondary hyperparathyroidism (those who received calcimimetics and calcium supplementation) in the 6 months leading up to paricalcitol treatment and during 6 months of paricalcitol treatment were also collected.
Time Frame: 6 months prior to start of study through 6 months of treatment
Population: This outcome measure was not analyzed due to lack of data.
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Hypercalcaemia During Preceding 6 Months of Conventional Vitamin D Therapy
Description: Hypercalcaemia (serum calcium > 2.6 mmol/L) among participants during the preceding 6 months of conventional vitamin D therapy was derived from retrospective data collection in case report form, reported at baseline. Conventional vitamin D therapy included vitamin D supplement products from ATC group A11CC (vitamin D and analogues).
Time Frame: 6 months prior to start of study through baseline
Population: Participants with available retrospective data
Measure: Number; unit: participants
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 58
participants | 5

7. Secondary Outcome: Number of Participants With Hypercalcaemia During 6 Months of Selective Vitamin D Receptor Activator (Paricalcitol) Treatment
Description: Hypercalcaemia (serum calcium > 2.6 mmol/L), based on laboratory data, was collected during the observed 6 months treatment with Zemplar (paricalcitol injection).
Time Frame: 6 months
Population: Participants with available retrospective data (cohort analyzed for Outcome Measure 6) were analyzed prospectively at Month 6 of treatment.
Measure: Number; unit: participants
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 58
participants | 20

8. Secondary Outcome: Number of Participants With Hyperphosphataemia During Preceding Conventional Vitamin D Therapy
Description: Hyperphosphataemia (serum phosphorus >1.78 mmol/L) among participants during the preceding 6 months of conventional vitamin D therapy was derived from retrospective data collection in case report form, reported at baseline. Conventional vitamin D therapy included vitamin D supplement products from ATC group A11CC (vitamin D and analogues).
Time Frame: 6 months prior to start of study through baseline
Population: Participants with available retrospective data
Measure: Number; unit: participants
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 54
participants | 39

9. Secondary Outcome: Number of Participants With Hyperphosphataemia During 6 Months of Selective Vitamin D Receptor Activator (Paricalcitol) Treatment
Description: Hyperphosphataemia (serum phosphorus > 1.78 mmol/L), based on laboratory data, was collected during the observed 6 months treatment with Zemplar (paricalcitol injection).
Time Frame: 6 months
Population: Participants with available retrospective data (cohort analyzed for Outcome Measure 8) were analyzed prospectively at Month 6 of treatment.
Measure: Number; unit: participants
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Number analyzed (Participants) | 54
participants | 50

ADVERSE EVENTS:
Time Frame: Reported from informed consent until 30 days or 5 half-lives following intake of last dose of physician-prescribed treatment. Thus, for each participant adverse events were assessed for a maximum of 7 months after the initial dose of Zemplar®.
Arm/Group | End-stage Kidney Disease With Secondary Hyperparathyroidism
Serious Adverse Events (participants affected / at risk) | 9/60
Other Adverse Events (participants affected / at risk) | 16/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | End-stage Kidney Disease With Secondary Hyperparathyroidism (N=60)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Inflammation (General disorders) | 1
Pyrexia (General disorders) | 1
Spinal pain (General disorders) | 1
Abscess limb (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (General disorders) | 1
Erysipelas (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Arterial occlusive disease (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | End-stage Kidney Disease With Secondary Hyperparathyroidism (N=60)
Calcium phosphate product increased (Investigations) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 7
Hyperphoshataemia (Metabolism and nutrition disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.